CLINICAL TRIAL: NCT07070349
Title: A Phase I/II Clinical Study to Evaluate the Safety, Radiation Dosimetry, Pharmacokinetics, and Preliminary Diagnostic Efficacy of HRS-6213 in Healthy Subjects and Patients With Solid Tumors
Brief Title: A Trial of HRS-6213 in Healthy Subjects and Patients With Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HRS-6213-101
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Patients With Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-6213 (Experimental)
  Interventions: Drug: HRS-6213

INTERVENTIONS:
Drug: HRS-6213 — HRS-6213 IV administered as imaging agent for PET scan.

SUMMARY:
The study is being conducted to evaluate the safety, radiation dosimetry, pharmacokinetics, and preliminary diagnostic efficacy of HRS-6213.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form; willing and able to follow the study protocol.
2. For healthy subjects：BMI 18~28kg/m2
3. For patients：

   * ECOG 0-1
   * Patients with pathologically confirmed tumour
   * proposed surgical resection/exploration (including primary or recurrent metastatic tumour
   * sufficient organs function.

Exclusion Criteria:

1. Known severe allergic reactions, hypersensitivity or contraindications to the test drug or any component of its preparation, such as alcohol allergy or other allergic history that the investigator deems may increase the risk of the trial.
2. Received the following treatments before administration:

   1. Received radionuclide diagnostic or therapeutic drugs before administration, and less than 10 physical half-lives have elapsed since the last administration.
   2. Used any intravenous iodinated contrast agent within 24 hours before administration, or used any high-density oral contrast agent within 5 days before administration (oral water-based contrast agent is acceptable).
3. Concurrent infectious diseases
4. Severe urinary incontinence, hydronephrosis, severe micturition dysfunction.
5. Concurrent severe active infection requiring intravenous antibiotic treatment within 14 days before administration.
6. Unexplained fever > 38.5℃ lasting for more than 1 hour during screening or before administration.
7. Concurrent severe or poorly controlled cardiac diseases or symptoms, including but not limited to: NYHA class 2 or higher heart failure, unstable angina, myocardial infarction within 6 months before administration, QTcF > 450 msec in males or QTcF > 470 msec in females.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Incidence of adverse events (AEs) of HRS-6213 | From first dose of study drug to end of treatment (up to approximately 7 days)
  To evaluate the safety and tolerability of HRS-6213.
Phase 1: Radiation dosimetry | From first dose of study drug to end of treatment (up to approximately 7 days)
  To evaluate the distribution of radioactivity in tissues and organs, and obtain the accumulation in major organs, time-radioactivity curves, internal radiation absorbed doses of the whole body and major organs of HRS-6213
Phase 2: With reference to the Standard of Truth (SOT), evaluate the diagnostic efficacy indicators of HRS-6213 PET at the lesion level | rom first dose of study drug to end of treatment (up to approximately 60 days)
  evaluate the diagnostic efficacy indicators of HRS-6213.

SECONDARY OUTCOMES:
Phase 1: Cmax | From first dose of study drug to end of treatment (up to approximately 7 days)
  To evaluate the PK of HRS-6213
Phase 1: Biological half-life (t½) | From first dose of study drug to end of treatment (up to approximately 7 days)
  To evaluate the PK of HRS-6213
Phase 1: Tmax | From first dose of study drug to end of treatment (up to approximately 7 days)
  To evaluate the PK of HRS-6213
Phase 1: urinary cumulative excretion rate | From first dose of study drug to end of treatment (up to approximately 7 days)
  To evaluate the PK of HRS-6213
Phase 1: Lesion uptake curve | From first dose of study drug to end of treatment (up to approximately 7 days)
  Lesion uptake curve of lesions detected by PET scans at different time points HRS-6213.
Phase 1: Image quality score | From first dose of study drug to end of treatment (up to approximately 7 days)
  Imaging quality scores of HRS-6213 with Likert image quality rating scale and signal-to-noise ratio.
Phase 2: The proportion of subjects with changes in disease staging and treatment decisions before and after HRS-6213 PET imaging. | From first dose of study drug to end of treatment (up to approximately 60 days)
  changes in disease staging and treatment decisions due to diagnostic test.
Phase 2: Intra-observer consistency of the diagnosticians' results | From first dose of study drug to end of treatment (up to approximately 7 days)
  consistency of the diagnosticians' results by investigators.
Phase 2:Incidence of adverse events (AEs) of HRS-6213 | From first dose of study drug to end of treatment (up to approximately 7 days)
  To evaluate the safety and tolerability of HRS-6213.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided